CLINICAL TRIAL: NCT04032041
Title: SCANREP: Reliability of 3D Lower Limb Scanning
Status: Terminated | Type: Observational
Why Stopped: No participants were enrolled for group 2. Study related activities were delayed due to the COVID pandemic and then terminated to focus on higher priority efforts.
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jason Wilken, Principal Investigator, University of Iowa
Other Study IDs: 201905871
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Foot Injuries and Disorders
Keywords: Ankle Foot Orthosis; Adult; 3D Limb Scanning; Limb Geometry
MeSH Terms: conditions — Foot Injuries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1: Healthy Able-bodied Individuals: Healthy able-bodied individuals with no history of lower extremity trauma.
  Interventions: Device: Structure Sensor; Device: Caliper
- Group 2: Individuals Requiring AFO Use: Individuals with unilateral, below knee functional deficits that require an AFO for daily activities (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease).
  Interventions: Device: Structure Sensor; Device: Caliper

INTERVENTIONS:
Device: Structure Sensor — A 3D representation of each participant's lower limb geometry will be obtained using a Structure Core scanner (Occipital, Inc.) which uses an infrared structured light projector to construct a 3D image of an object. The scanner is connected to an iPad; to operate the user rotates the iPad camera around the desired object. In seconds, the entire geometry is digitally reconstructed.
Device: Caliper — Caliper: An OriginCal IP54 digital caliper (Anytime Inc, Granada Hills, CA) was used to take three consecutive physical measurements in millimeters at each identified measurement location. For measurements outside of the caliper's scope a tape measure was used in place of the caliper. Physical measuring devices were reset to zero between each measure.

SUMMARY:
3D limb scanning systems have recently been implemented for the clinical fitting of prosthetic and orthotic devices due to substantial decreases in costs. However, little data is available regarding the repeatability and validity of systems currently in use. In this study the investigators seek to evaluate the repeatability and validity of multiple lower limb measurements obtained using low-cost 3D limb scanning technology.

DETAILED DESCRIPTION:
Two groups of subjects will be recruited for this study. The first group (Group 1) will consist of healthy able-bodied individuals with no history of lower extremity trauma. The second group (Group 2) will consist of individuals with unilateral, below knee functional deficits that require an AFO (ankle foot orthosis) for daily activities (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease).

The investigators will obtain a brief medical history to identify major medical conditions or prior injuries that could influence limb geometry, and lead to reliance on an AFO for Group 2 participants.

A 3D representation of each participant's lower limb geometry will be obtained using a Structure Core scanner (Occipital, Inc.) which uses an infrared structured light projector to construct a 3D image of an object. The scanner is connected to an iPad; to operate the user rotates the iPad camera around the desired object. In seconds, the entire geometry is digitally reconstructed. Measurements will be evaluated using digital imaging analysis software (Standard Cyborg, Inc.). The investigators will evaluate concurrent validity by directly comparing software-based measurements from limb scans, with direct measurements on the same individual collected using digital calipers. The investigators will determine repeatability of each technique by conducting three identical limb scans and actual physical measurements at two time points on the same day in each individual, and then comparing the results between time points. The interior of the AFO worn by participants in Group 2 will also be scanned to obtain its geometry for comparison with measurements obtained from each individual's limb.

Validity and repeatability will be assessed using measurements at multiple locations on the lower leg. Limb measurements will include 1) width of the metatarsal heads, 2) width of the calcaneus, 3) foot length, 4) foot height, 5) arch height, 6) medial-lateral width between ankle malleoli, 7) minimum circumference above the ankle malleoli, 8) maximum calf circumference , 9) medial-lateral width of the knee condyles 10) anterior-posterior width at mid patellar tendon, 11) distance from bottom of foot to tibial tubercle.

Concurrent validity will be determined using the intra-class correlation coefficient and absolute error (root mean square error) for comparisons between measurements from limb scanning and the calipers. Reliability will be determined using the intra-class correlation coefficient and the minimal detectable change value for comparisons over time.

ELIGIBILITY:
GROUP 1

Patient Inclusion criteria

* Ages: 18-75
* Healthy individuals without a current complaint of lower extremity pain, spine pain, active infections or medical or neuromusculoskeletal disorders that have limited participation in work or exercise in the last 6 months
* Ability to perform a full squat without pain
* Able to read and write in English and provide written informed consent

Patient Exclusion criteria

* Diagnosed moderate or severe brain injury
* Diagnosis of a physical or psychological condition that would preclude testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Current complaint of pain or numbness in the spine
* Uncorrected visual or hearing impairments that limit the ability to understand or comply with instructions given during testing
* Require an assistive device
* Open/unhealed wounds on lower extremity.
* BMI greater than 35

GROUP 2

Patient Inclusion criteria

* Ages: 18-75
* Daily AFO use to address unilateral below knee functional deficits (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease)
* Ability to stand independently without use of an assistive device (Cane, crutch, etc)
* Ability to safely bear full body weight on affected limb without use of an AFO or other protection
* Able to read and write in English and provide written informed consent

Patient Exclusion criteria

* Use of an AFO that crosses the knee (includes Knee brace or similar)
* Open/unhealed wounds on lower extremity
* Uncorrected visual or hearing impairments that limit the ability to understand or comply with instructions given during testing
* BMI greater than 35
* Diagnoses of a moderate to severe brain injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of subjects will be recruited for this study. The first group (Group 1) will consist of healthy able-bodied individuals with no history of lower extremity trauma. The second group (Group 2) will consist of individuals with unilateral, below knee functional deficits that require an AFO for daily activities (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participants were enrolled for group 2 (individuals requiring AFO use). Study related activities were delayed due to the COVID pandemic and then terminated to focus on higher priority efforts.
Groups:
- Group 1: Healthy Able-Bodied Individuals: Healthy able-bodied individuals with no history of traumatic lower limb injury.
  Caliper: An OriginCal IP54 digital caliper (Anytime Inc, Granada Hills, CA) was used to take three consecutive physical measurements in millimeters at each identified measurement location. For measurements outside of the caliper's scope a tape measure was used in place of the caliper. Physical measuring devices were reset to zero between each measure.
  Scan: A 3D representation of each participant's lower limb geometry will be obtained using a Structure Core scanner (Occipital, Inc.) which uses an infrared structured light projector to construct a 3D image of an object. The scanner is connected to an iPad; to operate the user rotates the iPad camera around the desired object. In seconds, the entire geometry is digitally reconstructed.
- Group 2: Individuals Requiring AFO Use: Individuals with unilateral, below knee functional deficits that require an AFO for daily activities (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease).
  Caliper: An OriginCal IP54 digital caliper (Anytime Inc, Granada Hills, CA) was used to take three consecutive physical measurements in millimeters at each identified measurement location. For measurements outside of the caliper's scope a tape measure was used in place of the caliper. Physical measuring devices were reset to zero between each measure.
  Scan: A 3D representation of each participant's lower limb geometry will be obtained using a Structure Core scanner (Occipital, Inc.) which uses an infrared structured light projector to construct a 3D image of an object. The scanner is connected to an iPad; to operate the user rotates the iPad camera around the desired object. In seconds, the entire geometry is digitally reconstructed.
Period: Overall Study
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Started | 30 | 0
Completed | 30 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled for group 2 (individuals requiring AFO use). Study related activities were delayed due to the COVID pandemic and then terminated to focus on higher priority efforts.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use | Total
Number analyzed (Participants) | 30 | 0 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 0 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (16) |  | 34.9 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 |  | 17
  Male | 13 |  | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Width of the Metatarsal Heads (Minimal Detectable Change [MDC])
Description: The width of the metatarsal heads was measured as the distance from the medial aspect of the first metatarsal head to the lateral aspect of the fifth metatarsal head. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intrarater-intersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper intrarater intersession | 1.1 |
  Scan intrarater intersession | 2.8 |
  Scan interrater intrasession | 2.2 |
  Scan interrater intersession | 3.1 |

2. Primary Outcome: Width of the Metatarsal Heads (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the width of the metatarsal heads. The width of the metatarsal heads is the distance from the medial aspect of the first metatarsal head to the lateral aspect of the fifth metatarsal head.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: Pearson's correlation coefficient values were calculated to compare between caliper and scan measurements. Pearson product-moment correlations were categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation.
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | 0.93 |

3. Primary Outcome: Width of the Metatarsal Heads (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the width of the metatarsal heads. The width of the metatarsal heads is the distance from the medial aspect of the first metatarsal head to the lateral aspect of the fifth metatarsal head.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 2.4 |

4. Primary Outcome: Width of the Calcaneus (Minimal Detectable Change [MDC])
Description: The width of the calcaneus was measured as the distance from the medial aspect of calcaneus parallel to lateral aspect of calcaneus. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper intrarater intersession | 0.8 |
  Scan intrarater intersession | 2.8 |
  Scan interrater intrasession | 1.1 |
  Scan interrater intersession | 3.0 |

5. Primary Outcome: Width of the Calcaneus (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the width of the calcaneus. The width of the calcaneus is the distance from the medial aspect of calcaneus parallel to lateral aspect of calcaneus.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | 0.93 |

6. Primary Outcome: Width of the Calcaneus (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the width of the calcaneus. The width of the calcaneus is the distance from the medial aspect of calcaneus parallel to lateral aspect of calcaneus.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 4.2 |

7. Primary Outcome: Foot Length (Minimal Detectable Change [MDC])
Description: Foot length was measured as the distance from the most posterior aspect of calcaneus to the most anterior toe (1st or 2nd). Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper intrarater intersession | 1.5 |
  Scan intrarater intersession | 3.2 |
  Scan interrater intrasession | 2.3 |
  Scan interrater intersession | 4.3 |

8. Primary Outcome: Foot Length (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the foot length. The foot length is the distance from the the most posterior aspect of calcaneus to the most anterior toe (1st or 2nd).
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | .99 |

9. Primary Outcome: Foot Length (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the foot length. The foot length is the distance from the most posterior aspect of calcaneus to the most anterior toe (1st or 2nd).
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 3.0 |

10. Primary Outcome: Foot Height (Minimal Detectable Change [MDC])
Description: Foot height was measured as the distance from the most superior point on the foot distal to the tibialis anterior insertion. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper Intrarater intersession | 2.1 |
  Scan intrarater intersession | 2.8 |
  Scan Interrater intrasession | 4.9 |
  Scan Interrater intersession | 5.9 |

11. Primary Outcome: Foot Height (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the foot height. The foot height is the distance from the most superior point on the foot distal to the tibialis anterior insertion.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | .8 |

12. Primary Outcome: Foot Height (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the foot height. The foot height is the distance from the most superior point on the foot distal to the tibialis anterior insertion.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 3.4 |

13. Primary Outcome: Arch Height (Minimal Detectable Change [MDC])
Description: Arch height was measured as the dorsum height at 50% foot length. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper Intrarater intersession | 2.3 |
  Scan intrarater intersession | 3.6 |
  Scan Interrater intrasession | 3.4 |
  Scan Interrater intersession | 5.8 |

14. Primary Outcome: Arch Height (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the arch height. The arch height is at 50% foot length.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | .85 |

15. Primary Outcome: Arch Height (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the arch height. The arch height is at 50% foot length.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 3.2 |

16. Primary Outcome: Medial-lateral Ankle Malleoli Width (Minimal Detectable Change [MDC])
Description: Medial-lateral ankle malleoli width was measured as the distance from the lateral malleolus to the medial malleolus. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper Intrarater intersession | 1.0 |
  Scan intrarater intersession | 2.6 |
  Scan Interrater intrasession | 1.2 |
  Scan Interrater intersession | 2.7 |

17. Primary Outcome: Medial-lateral Ankle Malleoli Width (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the width of the medial-lateral ankle malleoli. The width of the medial-lateral ankle malleoli is the distance from the lateral malleolus to the medial malleolus.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | .87 |

18. Primary Outcome: Medial-lateral Ankle Malleoli Width (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the width of the medial-lateral ankle malleoli. The width of the medial-lateral ankle malleoli is the distance from the lateral malleolus to the medial malleolus.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 2.8 |

19. Primary Outcome: Minimum Ankle Circumference (Minimal Detectable Change [MDC])
Description: Minimum ankle circumference was measured as the minimum ankle circumference above the ankle malleoli. Must be less than 10 cm proximal to the ankle malleoli. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper Intrarater intersession | 1.4 |
  Scan intrarater intersession MDC Scan intrarater intersession | 7.5 |
  Scan Interrater intrasession | 1.6 |
  Scan Interrater intersession | 8.1 |

20. Primary Outcome: Minimum Ankle Circumference (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the minimum ankle circumference. The minimum ankle circumference is the circumference above the ankle malleoli. Must be less than 10 cm proximal to the ankle malleoli.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | 0.93 |

21. Primary Outcome: Minimum Ankle Circumference (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the minimum ankle circumference. The minimum ankle circumference is the circumference above the ankle malleoli. Must be less than 10 cm proximal to the ankle malleoli.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 8.7 |

22. Primary Outcome: Maximum Calf Circumference (Minimal Detectable Change [MDC])
Description: Maximum calf circumference was measured as the maximum calf circumference greater that 5 cm distal to the knee condyles. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper Intrarater intersession | 4.3 |
  Scan intrarater intersession | 5.4 |
  Scan Interrater intrasession | 2.2 |
  Scan Interrater intersession | 5.8 |

23. Primary Outcome: Maximum Calf Circumference (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the maximum calf circumference. The maximum calf circumference is the distance greater than 5 cm distal to the knee condyles.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | .96 |

24. Primary Outcome: Maximum Calf Circumference (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the maximum calf circumference. The maximum calf circumference is the distance greater than 5 cm distal to the knee condyles.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 7.2 |

25. Primary Outcome: Width of the Knee Condyles (Minimal Detectable Change [MDC])
Description: Width of the knee condyles was measured as the distance from the medial condyle to the lateral condyle. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper Intrarater intersession | 3.4 |
  Scan intrarater intersession | 4.2 |
  Scan Interrater intrasession | 1.4 |
  Scan Interrater intersession | 4.2 |

26. Primary Outcome: Width of the Knee Condyles (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for the width of the knee condyles. The width of the knee condyles is the distance from the medial condyle to the lateral condyle.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | .98 |

27. Primary Outcome: Width of the Knee Condyles (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the width of the knee condyles. The width of the knee condyles is the distance from the medial condyle to the lateral condyle.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 3.9 |

28. Primary Outcome: Anterior-posterior Width at Patella (Minimal Detectable Change [MDC])
Description: Anterior-posterior width at patella was measured as the distance from mid patellar tendon to a parallel point most posterior on the back of the knee. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper Intrarater intersession | 4.8 |
  Scan intrarater intersession | 3.7 |
  Scan Interrater intrasession | 1.5 |
  Scan Interrater intersession | 3.7 |

29. Primary Outcome: Anterior-posterior Width at Patella (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated for anterior-posterior width at patella. The anterior-posterior width at patella is the distance from mid patellar tendon to a parallel point most posterior on the back of the knee.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | 0.93 |

30. Primary Outcome: Anterior-posterior Width at Patella (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for anterior-posterior width at patella. The anterior-posterior width at patella is the distance from mid patellar tendon to a parallel point most posterior on the back of the knee.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 6.0 |

31. Primary Outcome: Tibial Tubercle Height (Minimal Detectable Change [MDC])
Description: Tibial tubercle height was measured as the distance from the floor to tibial tubercle. Reliability of these measures was assessed using minimal detectable change (MDC) values. MDC values are in the same units as the original measure, and smaller values are better. Minimal Detectable Change (MDC) values are presented for: caliper intraraterintersession, scan intrarater-intersession, scan interrater-intrasession, and scan interrater-intersession.
  MDCs were calculated for all participants as a whole using the equation SEM x 1.96 x SQRT where SEM was calculated using the equation SD x SQRT (1-ICC), where SD is the pooled variance. ICC values were calculated using SPSS v.25 using model (2,k). [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for baseline characteristics
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Caliper Intrarater intersession | 3.6 |
  Scan intrarater intersession | 5.2 |
  Scan Interrater intrasession | 6.3 |
  Scan Interrater intersession | 7.9 |

32. Primary Outcome: Tibial Tubercle Height (Pearson's Correlation Coefficient)
Description: Pearson's correlation coefficient was calculated tibial tubercle height. The tibial tubercle height is the distance from the floor to tibial tubercle.
  Pearson product-moment correlations were calculated for all participants as a whole to compare between caliper and scan measurements using the function PEARSON (array1, array2) and categorized based on the scale of negligible (0-0.30), low (0.30-0.50), moderate (0.50-0.70), high (0.70-0.90), and very high (0.90-1.0) correlation. [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
correlation coefficient | .97 |

33. Primary Outcome: Tibial Tubercle Height (Mean Root Mean Square [RMS] Difference)
Description: The mean Root Mean Square (RMS) difference was calculated for the tibial tubercle height. The tibial tubercle height is the distance from the floor to tibial tubercle.
  RMS was calculated by squaring the mean for all participants, adding up the squares (which are all positive) and dividing by the number of samples to find the average square or mean square, then taking the square root of that. And the root mean square difference was calculated by comparing caliper and scan measurements [Powers OA, et al. (2022), Prosthet Orthot Int. 46(1)]
  Data is only presented for group 1 as study activities related to group 2 were terminated due to the COVID pandemic.
Time Frame: Less than 2 days
Population: RMS difference values were calculated to compare between caliper and scan measurements.
Measure: Number; unit: mm
Arm/Group | Group 1: Healthy Able-Bodied Individuals | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm | 5.8 |

34. Primary Outcome: Bland-Altman Plots
Description: Bland-Altman plot (difference plot) is a method of data plotting used in analyzing the agreement between scan and caliper measures for each identified measurements.
Time Frame: Less than 2 days
Population: No participants were enrolled for group 2. Study related activities were delayed due to the COVID pandemic and then terminated to focus on higher priority efforts.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Group 1: Healthy Able-bodied Individuals (Completed): Healthy able-bodied individuals with no history of lower extremity trauma.
  Structure Sensor: A 3D representation of each participant's lower limb geometry will be obtained using a Structure Core scanner (Occipital, Inc.) which uses an infrared structured light projector to construct a 3D image of an object. The scanner is connected to an iPad; to operate the user rotates the iPad camera around the desired object. In seconds, the entire geometry is digitally reconstructed.
Arm/Group | Group 1: Healthy Able-bodied Individuals (Completed) | Group 2: Individuals Requiring AFO Use
Number analyzed (Participants) | 30 | 0
mm
  Width of metatarsal heads | -0.09 (1.68) |
  Width of calcaneus | -3.50 (2.21) |
  Foot height | 1.16 (2.49) |
  Medial arch height | 1.01 (2.14) |
  Medial-lateral width between ankle malleoli | -1.59 (1.68) |
  Foot length | -1.37 (1.73) |
  Minimum circumference above the ankle malleoli | -5.78 (5.73) |
  Maximum calf circumference | -2.14 (4.13) |
  Medial-lateral width of the knee condyles | -2.99 (2.27) |
  Anterior-posterior width at mid patellar tendon | -4.46 (3.23) |
  Distance from bottom of foot to tibial tubercle | -1.41 (3.99) |

35. Primary Outcome: Intrarater-intersession ICC Values
Description: Intrarater-intersession ICC values were calculated to determine the test-retest reliability of scanning and digital measurements, whereas inter-rater-intrasession and inter-rater-intersession ICC values were calculated to determine the reliability of digital measurements. Intrarater-intersession ICC values were calculated to determine the reliability of physical measures between sessions. ICC values generally range from 0-1 with higher values indicating better reliability
Time Frame: Less than 2 days
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Caliper Intrarater-intersession; Scan Intrarater-intersession; Scan Inter-rater-intrasession; Scan Inter-rater Intersession: Healthy able-bodied individuals with no history of lower extremity trauma.
Arm/Group | Caliper Intrarater-intersession | Scan Intrarater-intersession | Scan Inter-rater-intrasession | Scan Inter-rater Intersession
Number analyzed (Participants) | 30 | 30 | 30 | 30
correlation coefficient
  Width of metatarsal heads | 0.99 [0.99 to 0.99] | 0.98 [0.95 to 0.99] | 0.99 [0.97 to 0.99] | 0.97 [0.94 to 0.99]
  Width of calcaneus | 0.99 [0.99 to 1.00] | 0.98 [0.95 to 0.99] | 0.99 [0.99 to 0.99] | 0.97 [0.94 to 0.99]
  Foot height | 0.97 [0.94 to 0.99] | 0.97 [0.93 to 0.98] | 0.89 [0.77 to 0.95] | 0.84 [0.67 to 0.92]
  Arch height | 0.98 [0.96 to 0.99] | 0.94 [0.88 to 0.97] | 0.95 [0.90 to 0.98] | 0.85 [0.68 to 0.93]
  Medial-lateral width between ankle malleoli | 0.99 [0.99 to 1.00] | 0.96 [0.92 to 0.98] | 0.99 [0.98 to 0.99] | 0.96 [0.91 to 0.98]
  Foot length | 0.99 [0.99 to 1.00] | 0.99 [0.99 to 1.00] | 0.99 [0.99 to 1.00] | 0.99 [0.98 to 0.99]
  Minimum circumference above the ankle malleoli | 0.99 [0.99 to 1.00] | 0.98 [0.95 to 0.99] | 0.99 [0.99 to 1.00] | 0.97 [0.94 to 0.99]
  Maximum calf circumference | 0.99 [0.99 to 1.00] | 0.99 [0.98 to 0.99] | 1.00 [0.99 to 1.00] | 0.99 [0.98 to 0.99]
  Medial-lateral width of the knee condyles | 0.99 [0.97 to 0.99] | 0.98 [0.96 to 0.99] | 0.99 [0.99 to 1.00] | 0.98 [0.96 to 0.99]
  Anterior-posterior width at mid patellar tendon | 0.96 [0.92 to 0.98] | 0.98 [0.96 to 0.99] | 0.99 [0.99 to 1.00] | 0.98 [0.96 to 0.99]
  Distance from bottom of foot to tibial tubercle | 0.99 [0.99 to 1.00] | 0.99 [0.99 to 1.00] | 0.99 [0.98 to 0.99] | 0.99 [0.97 to 0.99]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed before starting study activities and after each round of measurement (caliper/scan) during the study visit (~1 hour). Monitoring stopped at the end of the study visit but participants were instructed to contact the research team and report adverse events following the study visit, up to a maximum of 12 months post study completion.
Description: No participants were enrolled for group 2 (individuals requiring AFO use). Study related activities were delayed due to the COVID pandemic and then terminated to focus on higher priority efforts. Therefore, the number of participants at risk for group 2 is zero.
Groups:
- Group 2: Individuals Requiring AFO Use (Completed): Individuals with unilateral, below knee functional deficits that require an AFO for daily activities (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease).
  Structure Sensor: A 3D representation of each participant's lower limb geometry will be obtained using a Structure Core scanner (Occipital, Inc.) which uses an infrared structured light projector to construct a 3D image of an object. The scanner is connected to an iPad; to operate the user rotates the iPad camera around the desired object. In seconds, the entire geometry is digitally reconstructed.
Arm/Group | Group 1: Healthy Able-bodied Individuals (Completed) | Group 2: Individuals Requiring AFO Use (Completed)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/0
Other Adverse Events (participants affected / at risk) | 0/30 | 0/0

LIMITATIONS AND CAVEATS:
No participants were enrolled for group 2 (individuals requiring AFO use). Study related activities were delayed due to the COVID pandemic and then terminated to focus on higher priority efforts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04032041/Prot_SAP_000.pdf